CLINICAL TRIAL: NCT06375720
Title: Dose-effect of Different Frequencies and Duration of Tai Chi Chuan to Improve Cognitive Function in Persons With Mild Cognitive Impairment
Brief Title: Efficacy of Different Doses of Tai Chi Chuan on Cognitive Function in Persons With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lidian Chen (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor-Investigator, Lidian Chen, Fujian University of Traditional Chinese Medicine, Fujian University of Traditional Chinese Medicine
Organization: Fujian University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FujianUTCM-2
Record Dates: First submitted 2024-03-21; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Tai Chi Chuan; Cognitive Function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Tai Chi Chuan Group1 (Experimental): 12 weeks of Tai Chi Chuan, 3x/week
  Interventions: Behavioral: Lower frequency, shorter period of Tai Chi Chuan
- Tai Chi Chuan Group2 (Experimental): 12 weeks of Tai Chi Chuan, 5x/week
  Interventions: Behavioral: Higher frequency, shorter period of Tai Chi Chuan
- Tai Chi Chuan Group3 (Experimental): 24 weeks of Tai Chi Chuan, 3x/week
  Interventions: Behavioral: Lower frequency, longer period of Tai Chi Chuan
- Tai Chi Chuan Group4 (Experimental): 24 weeks of Tai Chi Chuan, 5x/week
  Interventions: Behavioral: Higher frequency, longer period of Tai Chi Chuan
- Control (Sham Comparator): Participants would take standard health education 0.5hour/ session, 2 sessions/month for 6 months.
  Interventions: Behavioral: Standard Health Education

INTERVENTIONS:
Behavioral: Lower frequency, shorter period of Tai Chi Chuan — Participants would take 24-form simplified Tai Chi Chuan 1 hour/session, 3 sessions/week for 12 weeks. There were 10 minutes warm-up, 40 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training. Besides, they would also take standard health education 0.5 hour/session, 2 sessions/month for 6 months.
  Arms: Tai Chi Chuan Group1
Behavioral: Higher frequency, shorter period of Tai Chi Chuan — Participants would take 24-form simplified Tai Chi Chuan 1 hour/session, 5 sessions/week for 12 weeks. There were 10 minutes warm-up, 40 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training. Besides, they would also take standard health education 0.5 hour/session, 2 sessions/month for 6 months.
  Arms: Tai Chi Chuan Group2
Behavioral: Lower frequency, longer period of Tai Chi Chuan — Participants would take 24-form simplified Tai Chi Chuan 1 hour/session, 3 sessions/week for 24 weeks. There were 10 minutes warm-up, 40 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training. Besides, they would also take standard health education 0.5 hour/session, 2 sessions/month for 6 months.
  Arms: Tai Chi Chuan Group3
Behavioral: Higher frequency, longer period of Tai Chi Chuan — Participants would take 24-form simplified Tai Chi Chuan 1 hour/session, 5 sessions/week for 24 weeks. There were 10 minutes warm-up, 40 minutes Tai Chi Chuan lesson and 10 minutes cool-down exercises in the Tai Chi Chuan training. Besides, they would also take standard health education 0.5 hour/session, 2 sessions/month for 6 months.
  Arms: Tai Chi Chuan Group4
Behavioral: Standard Health Education — Participants would take standard health education 0.5 hour/ session, 2 sessions/month for 6 months.
  Arms: Control

SUMMARY:
To determine the relationship between the effects of different frequencies and duration of Tai Chi Chuan in dose parameters to improve cognitive function in elderly persons with mild cognitive impairment.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) is regarded as a prodrome to dementia and affects 16% to 20% of people aged older than 65 years. Tai Chi Chuan is an increasingly popular multi-modal physical and mental exercise. Studies have shown that Tai Chi Chuan can effectively improve the cognitive function of elderly persons with MCI. However, the relationship between the effects of different frequencies and duration of Tai Chi Chuan to improve the cognitive function of elderly persons with MCI is not yet clear. The purpose of this study is to determine the optimal frequency and duration of Tai Chi Chuan. The investigators will conduct a single-blind, randomized controlled trial in 350 persons who meet the presence of MCI without dementia. Persons will be randomly assigned to either the Tai Chi Chuan intervention group once or twice a week for 12 or 24 weeks, or the health education control group once every four weeks for 24 weeks. All groups will be followed for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of mild cognitive impairment, not demented;
2. Age ≥ 60 years old;
3. Informed consent and voluntary participation.

Exclusion Criteria:

1. Geriatric Depression Scale score ≥ 9 points;
2. Cognitive impairment caused by other reasons, taking drugs, poisoning, etc;
3. Suffer from severe musculoskeletal system diseases and other contraindications to exercise and are not suitable for Tai Chi Chuan training, such as those who suffer from stroke, Parkinson's disease, and have a history of lower limb arthritis, hip and knee joint replacement, etc;
4. Patients with severe heart, liver, kidney failure, malignant tumors, and other major diseases;
5. Individuals with visual/auditory impairments, writing/reading impairments, illiteracy, etc. that affect training and evaluation;
6. Individuals with uncontrolled hypertension (systolic blood pressure greater than 160mmHg or diastolic blood pressure greater than 100mmHg after medication);
7. Participating in other experiments that influence this study;
8. Engaged in regular exercise in the last three months (at least 3 times a week, at least 20 minutes of regular exercise each time).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-05-05 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | 12 weeks, 24 weeks
  Global cognition

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | 52 weeks
  Global cognition
Wechsler Memory Scale | 12 weeks, 24 weeks and 52 weeks
  Memory function
Digit Symbol Substitution Test | 12 weeks, 24 weeks and 52 weeks
  Attention
Trial Making Test part B | 12 weeks, 24 weeks and 52 weeks
  Executive Function
Stroop Color Word Test | 12 weeks, 24 weeks and 52 weeks
  Processing Speed
Boston Naming Test | 12 weeks, 24 weeks and 52 weeks
  Verbal fluency
Rey-Osterrieth Complex Graphics Test | 12 weeks, 24 weeks and 52 weeks
  Visuo-spatial ability
Rey Auditory Verbal Learning Test | 12 weeks, 24 weeks and 52 weeks
  Episodic memory

OTHER OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 12 weeks, 24 weeks and 52 weeks
  Sleep quality
12-Item Short Form Health Survey | 12 weeks, 24 weeks and 52 weeks
  General health
Blood glucose metabolism index | 12 weeks, 24 weeks and 52 weeks
  fasting blood glucose
Blood lipid metabolism index | 12 weeks, 24 weeks and 52 weeks
  total cholesterol (TC); total triglyceride (TG); low density lipoprotein (LDL);high density lipoprotein (HDL)
functional Magnetic Resonance Imaging | 12 weeks or 24 weeks [post-intervention]
  functional Magnetic Resonance Imaging
Electroencephalogram | 12 weeks or 24 weeks [post-intervention]
  The power spectrum density of the brain in a relaxed state is measured using a resting-state electroencephalogram (EEG) for the delta (1-4 Hz), theta (4-8 Hz), alpha (8-13 Hz), beta (13-30 Hz), and gamma (30-100 Hz) bands.
Heart rate variability | 12 weeks or 24 weeks [post-intervention]
  Cardiac autonomic modulations
Gut microflora | 12 weeks, 24 weeks and 52 weeks
  16S rRNA amplification sequencing was used to detect intestinal microbiota.